CLINICAL TRIAL: NCT00401570
Title: Phase 2 Open-Label Study of Volociximab (M200) in Combination With Gemcitabine in Patients With Metastatic Pancreatic Cancer Not Previously Treated With Chemotherapy
Brief Title: A Study of Volociximab in Combination With Gemcitabine in Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M200-1205
Record Dates: First submitted 2006-11-16; First posted 2006-11-20 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Pancreatic Cancer
Keywords: Antibody; Pancreas; Carcinoma; Cancer; Pancreatic
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma; Neoplasms | interventions — volociximab; Gemcitabine

ARMS (2):
- Cohort 1 (Experimental): Volociximab (10 mg/kg every other week (qowk)) and Gemcitabine
  Interventions: Drug: Volociximab; Drug: Gemcitabine
- Cohort 2 (Experimental): Volociximab (15 mg/kg weekly (qwk)) and Gemcitabine
  Interventions: Drug: Volociximab; Drug: Gemcitabine

INTERVENTIONS:
Drug: Volociximab — Volociximab: 10 mg/kg or 15mg/kg every week or every other week (qowk) via IV infusion for up to 104 weeks.
Drug: Gemcitabine — Gemcitabine: Standard chemotherapy regime at 1 g/m2 once per week for 3 weeks via IV infusion, followed by one week with no treatment

SUMMARY:
This clinical trial is being conducted to determine tumor response and preliminary safety of a monoclonal antibody that specifically binds to a cell surface receptor (α5β1 integrin) that is required for the establishment of new blood vessels during tumor growth, a process known as angiogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older.
* Histologically or cytologically confirmed metastatic adenocarcinoma of the pancreas.
* May have received prior immunotherapy (including monoclonal antibodies) or vaccine therapies.
* Measurable disease, according to RECIST criteria.
* Negative pregnancy test (women of childbearing potential only).
* Pretreatment laboratory levels that meet specific criteria.

Exclusion Criteria:

* Prior treatment with Volociximab (M200) or inhibitors of α5β1 integrin (antibodies or small molecules) or gemcitabine and other chemotherapeutic regimens.
* Known hypersensitivity to murine proteins or chimeric antibodies or other components of the product.
* Use of any investigational drug within 4 weeks prior to screening or 5 half-lives of the prior investigational drug (whichever is longer).
* Monoclonal antibody therapy within 4 weeks of the first dose of Volociximab.
* Central Nervous System (CNS) tumor or metastasis.
* History of bleeding disorders within the past year.
* Medical conditions that may be exacerbated by bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The proportion of patients, in each dose cohort, with a confirmed tumor response | Any time during the course of the trial (up to 104 weeks)

SECONDARY OUTCOMES:
Duration of progression-free survival | During the course of the trial (up to 104 weeks)
Time to disease progression | During the course of the trial (up to 104 weeks)
Duration of overall survival | During the course of the trial (up to 104 weeks)
To evaluate the safety in of M200 in combination with gemcitabine | During the course of the trial (up to 104 weeks)
To evaluate the pharmacokinetics of M200 | During the course of the trial (up to 104 weeks)
To evaluate the immunogenicity of M200 | During the course of the trial (up to 104 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Mihail Obrocea, MD, Study Director — AbbVie
Locations (6):
- United States (2):
  - Site Reference ID/Investigator# 70538, Pittsburgh, Pennsylvania
  - Site Reference ID/Investigator# 70537, Nashville, Tennessee
- United Kingdom (4):
  - Site Reference ID/Investigator# 70534, Glasgow
  - Site Reference ID/Investigator# 70533, Leeds
  - Site Reference ID/Investigator# 70536, Manchester
  - Site Reference ID/Investigator# 70535, Northwood